CLINICAL TRIAL: NCT01528683
Title: Phase I/II Trial Evaluating Carbon Ion Radiotherapy for the Treatment of Recurrent Rectal Cancer
Acronym: PANDORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANDORA
Record Dates: First submitted 2011-12-31; First posted 2012-02-08 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Recurrent Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbon Ion Radiotherapy (Experimental)
  Interventions: Radiation: Carbon Ion Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Treatment with carbon ion radiotherapy using the rasterscanning technique

SUMMARY:
Treatment standard for patients with rectal cancer depends on the initial staging and includes surgical resection, radiotherapy as well as chemotherapy. For stage II and III tumors, radiochemotherapy should be performed in addition to surgery, preferentially as preoperative radiochemotherapy or as short-course hypofractionated radiation. Advances in surgical approaches, especially the establishment of the total mesorectal excision (TME) in combination with sophisticated radiation and chemotherapy have reduced local recurrence rates to only few percent. However, due to the high incidence of rectal cancer, still a high absolute number of patients present with recurrent rectal carcinomas, and effective treatment is therefore needed.

Carbon ions offer physical and biological characteristics. Due to their inverted dose profile and the high local dose deposition within the Bragg peak precise dose application and sparing of normal tissue is possible. Moreover, in comparison to photons, carbon ions offer an increase relative biological effectiveness (RBE), which can be calculated between 2 and 5 depending on the cell line as well as the endpoint analyzed.

Japanese data on the treatment of patients with recurrent rectal cancer previously not treated with radiation therapy have shown local control rates of carbon ion treatment superior to those of surgery. Therefore, this treatment concept should also be evaluated for recurrences after radiotherapy, when dose application using conventional photons is limited. Moreover, these patients are likely to benefit from the enhanced biological efficacy of carbon ions.

In the current Phase I/II-PANDORA-01-Study the recommended dose of carbon ion radiotherapy for recurrent rectal cancer will be determined in the Phase I part, and feasibility and progression-free survival will be assessed in the Phase II part of the study.

Within the Phase I part, increasing doses from 12 x 3 Gy E to 18 x 3 Gy E will be applied.

The primary endpoint in the Phase I part is toxicity, the primary endpoint in the Phase II part its progression-free survival.

ELIGIBILITY:
Inclusion Criteria

* Locally recurrent rectal cancer
* Inoperable lesion
* Macroscopic tumor up to 1000ml volume- prior photon radiation of 20-60 Gy
* time between initial radiotherapy and re-irradiation of at least 12 months
* age ≥ 18 years of age
* Karnofsky Performance Score >60
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria

* refusal of the patients to take part in the study
* advanced metastatic disease
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy- Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy | 3 months
  Phase I part:
  The primary endpoint is toxicity measured by any Grade IV toxicity related to the study treatment according to CTCAE Grade 41. A maximum of 45 patients are projected for the Phase I part of the study. Patients will be followed for at least 3 months after study treatment to document any toxicity according to CTCAE Version 4.0.
  Phase II part:
  The primary endpoint is progression-free survival after re-irradiation at 12 months, therefore patients are followed within the trial protocol for a minimum 12 months after completion of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, MD PhD, Principal Investigator — University Hospital of Heidelberg
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Habermehl D, Wagner M, Ellerbrock M, Buchler MW, Jakel O, Debus J, Combs SE. Reirradiation Using Carbon Ions in Patients with Locally Recurrent Rectal Cancer at HIT: First Results. Ann Surg Oncol. 2015;22(6):2068-74. doi: 10.1245/s10434-014-4219-z. Epub 2014 Nov 11. PMID 25384705
- [Derived] Combs SE, Kieser M, Habermehl D, Weitz J, Jager D, Fossati P, Orrechia R, Engenhart-Cabillic R, Potter R, Dosanjh M, Jakel O, Buchler MW, Debus J. Phase I/II trial evaluating carbon ion radiotherapy for the treatment of recurrent rectal cancer: the PANDORA-01 trial. BMC Cancer. 2012 Apr 3;12:137. doi: 10.1186/1471-2407-12-137. PMID 22472035